CLINICAL TRIAL: NCT02826473
Title: Analysis of Clinical- and Cost-effectiveness of Focused Cognitive Testing in Elective Inpatients
Brief Title: Focused Cognitive Testing in Inpatients
Acronym: FCTI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment of eligible patients
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Universität Luzern (Other)
Responsible Party: Principal Investigator, Aljoscha Hwang, Health Research Manager, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LUKS-2016-00140; 2016-00140 (Other: Ethics Committee Northwest and Central Switzerland)
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Neurocognitive Disorders
Keywords: Dementia; Dementia screening; General Hospital; Inpatients
MeSH Terms: conditions — Neurocognitive Disorders; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Group (Experimental)
  Interventions: Other: BRAINCHECK
- Control-Group (No Intervention)

INTERVENTIONS:
Other: BRAINCHECK — Subjects of the Intervention-Group will undergo a brief cognitive assessment, using the BRAINCHECK, during hospital admission assessments. Subjects with positive results will then be referred to a Memory Clinic undergoing subsequent interdisciplinary comprehensive diagnostic examinations. Patients with established diagnosis will be invited to counselling services of the Alzheimer Association (providing social counselling).
  Arms: Intervention-Group

SUMMARY:
Neurocognitive Disorder (NCD) affects over 116'000 people in Switzerland and is frequently unrecognized and underdiagnosed. Because missed and delayed diagnosis are associated with an increased burden of disease health Service Research has prompted a discussion about diagnostic guidelines and screening programs. Some argue that screening for NCD in primary care is the optimal strategy to increase recognition rates; others consider test protocols implemented into hospital admission assessments as more justified. There is no distinct recommendation due to a lack of empirical data on the benefits and harms of cognitive testing yet. This trial strives to fill this gap and provide information about the benefits, harms and the economic case of routine cognitive testing for neurocognitive disorder in high risk elective inpatients, in Switzerland.

The investigators hypothesize that, cognitive tested patients, compared with patients not cognitive tested, will have higher health-related quality of life at 12months; and lower medical health care costs at 18months.

ELIGIBILITY:
Inclusion Criteria:

* Elective inpatients, living in the canton of lucerne, high risk of developing a major neurocognitive disorder, living at home

Exclusion Criteria:

* Known mental disorder according to ICD-10, chapter V, excluding F32 & F33, patients with terminal illness, patients of intensive care unit or oncology patients, no adequate vision or hearing, no ability to speak, write or to understand German, no Informant, antidementia medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (HRQoL) | every month during 18months
  Patient and Caregiver, using EuroQol 5D-5L
Health Service Resource Utilization / Costs | every month during 18months
  Patient and Caregiver, using Resource Utilization in Dementia (RUD)

SECONDARY OUTCOMES:
prevalence of neurocognitive disorder | baseline/6months
  at Hospital admission
prevalence of risk factors associated with developing major neurocognitive disorder within 6 years | baseline/6months
  at Hospital Admission, using Brief Dementia Screening Indicator (BDSI)

OTHER OUTCOMES:
caregiver burden | every 3 months
  caregiver data, short Zarit Burden Interview (ZBI)
adverse events/adverse outcomes | between baseline and 6months
  falls, delirium, mortality, mortality within 30 days of discharge, re-admission within 18 days, institutionalization following hospitalization, length of stay
comorbidities | baseline
  patient data, using Charlson Comorbidity Index
neuropsychiatric symptoms | between baseline and 6months
  patient data during Hospital stay, using Neuropsychiatric Inventory Questionnaire (NPI-Q)
hospital anxiety and depression | every 3 months
  patient and caregiver data, using Hospital Anxiety and Depression Scale (HADS)
severity of cognitive impairment | every 6 months
  patients of the Intervention-Group will be assessed every months, using the Montreal Cognitive Assessment (MOCA)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Boes, Prof.Dr., Principal Investigator — University of Lucerne,Department of Health Sciences & Health Policy; Thomas Nyffeler, Prof.Dr.med., Study Chair — Cantonal Hospital of Lucerne; Aljoscha Benjamin, M.A. (HSG), Study Chair — Cantonal Hospital of Lucerne
Locations (1):
- Cantonal Hospital of Lucerne, Lucerne, Canton Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No